CLINICAL TRIAL: NCT06951074
Title: Autologous Insulin Producing Mesenchymal Stem Cell Transplantation in Youth With Type 1 Diabetes
Brief Title: Insulin Producing Stem Cell Transplantation Clinical Trial in Type 1 Diabetes
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AinShamsPedDiabetes
Record Dates: First submitted 2025-04-04; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-01

CONDITIONS: Stem Cells; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Twenty youth with T1D, aged 15 to 18 years will participate in this clinical trial. The International Society for Pediatric and Adolescent Diabetes (ISPAD) guidelines for Type 1 diabetes diagnosis (2024) will be used to confirm the diagnosis of Type 1 Diabetes. Patients' group will be subsequently separated into two subgroups 1a and 1b, each of which contain 10 patients. Group 1a will represent patients who will receive the insulin producing MScs through the portal circulation via Ultrasound guided portal vein injection. Group 1b will represent the patients who will receive the insulin producing MScs through the systemic circulation via peripheral cannulation. The Pediatrics and Adolescent Diabetic Clinic at Ain Shams University Hospital will be used to enroll T1D participants. Patients involved in the study will be admitted in the Pediatric Hospital (El-Demerdash)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1a IPSC transplant in portal circulation (Experimental): Insulin producing stem cells injection in portal circulation
  Interventions: Biological: Insulin producing stem cells infusion
- group 1b IPSC in peripheral systemic circulation (Experimental): Insulin producing stem cells injection in peripheral systemic circulation
  Interventions: Biological: Insulin producing stem cells infusion

INTERVENTIONS:
Biological: Insulin producing stem cells infusion — 1. Liposuction of the anterior abdominal subcutaneous fat layer of participant
  2. Characterization and Identification of mesenchymal stem cells
  3. Differentiation of mesenchymal stem cells into insulin producing stem cells
  4. In vitro detection of Insulin and c-peptide in differentiated MSC (Confirmatory tests for the insulin producing cells)
  5. In vitro Insulin and c-peptide release detection in differentiated MSC in response to increasing glucose concentrations Differentiated MSCs injection in human subjects
  6. Followup

SUMMARY:
Type 1 Diabetes is a chronic autoimmune disease. It results from autoimmune destruction of pancreatic Beta cells leading to absolute insulin insufficiency. The establishment of pluripotent like human stem cells derived from adipose tissue derived mesenchymal cell origin have introduced a new potential source for cell therapy in type 1 diabetic patients, especially in light of recent successes in producing glucose-sensitive insulin secreting cells and this will be the scope of this study. In the last decade, human clinical trials of introducing insulin producing stem cells from various origins were approved and conducted.

DETAILED DESCRIPTION:
Differentiation of stem cells from various sources to form insulin-producing cells (IPCS) provides a new and promising strategy to reconstitute pancreatic endocrine function. Studies recently developed a multistep differentiation technique for the differentiation of human embryonic stem cells to form pancreatic progenitors. At the end of in vitro differentiation approximately 5% of cells became insulin positive.

Mesenchymal stem cells (MSCs) can be derived from various sources. MSCs are undifferentiated cells with multilinear potential, known for their immunomodulatory and regenerative properties . The bone marrow, adipose tissue, umbilical cord, liver cells, and endometrium are among several tissues that are rich in MSCs. Of these, the bone marrow and adipose tissues offer distinct advantages in view of their availability and abundance and the extent of their documentation.

In this study the investigators aim to obtain autologous differentiated insulin producing mesenchymal stem cells (derived from adipose tissue) and their introduction in human subjects with type 1 diabetes. The current study will assess of the ability of the transplanted cells to produce insulin both in vitro and in vivo. Post- transplant glycemic control will be assessed with possible amelioration of the standard treatment of type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes

Exclusion Criteria:

* patients with other autoimmune diseases
* patients with micro or macro vascular complications
* patients with other chronic diseases

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Insulin producing mesenchymal stem cells efficacy in insulin production in vitro | 1 year
  Assessment of the percentage of mature insulin and c peptide production in insulin producing stem cells.
Insulin producing mesenchymal stem cells efficacy in insulin production in vitro | 1 year
  Assestment of percentage of mature insulin production and c peptide in insulin producing stem cells in response to different concentrations of glucose.
Insulin producing mesenchymal stem cells efficacy in insulin production in vivo | 1 year
  Participants glycemic control will be assesed before and after insulin producing stem cells injection.

CONTACTS AND LOCATIONS:
Overall Officials: Rasha S Elmetwally, A. Prof, Principal Investigator — Assistant professor of Pediatrics, Faculty of Medicine, Ain Shams University; Randa M Matter, Prof, Study Director — Professor of pediatrics, Faculty of Medicine, Ain Shams University
Locations (1):
- Children Hospital Eldemerdash, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abou Zaki R, El-Osta A. Advancing type 1 diabetes therapy: autologous islet transplant breakthrough. Signal Transduct Target Ther. 2024 Dec 23;9(1):366. doi: 10.1038/s41392-024-02090-x. No abstract available. PMID 39710778
- [Background] Ulyanova O, Askarov M, Kozina L, Karibekov T, Shaimardanova G, Zhakupova A, Danilova D, Serebrennikova D. Autologous Mesenchymal Stem Cell Transplant in Patients with Type 1 Diabetes Mellitus. Exp Clin Transplant. 2019 Jan;17(Suppl 1):236-238. doi: 10.6002/ect.MESOT2018.P100. PMID 30777564
- [Background] Jayasinghe M, Prathiraja O, Perera PB, Jena R, Silva MS, Weerawarna PSH, Singhal M, Kayani AMA, Karnakoti S, Jain S. The Role of Mesenchymal Stem Cells in the Treatment of Type 1 Diabetes. Cureus. 2022 Jul 27;14(7):e27337. doi: 10.7759/cureus.27337. eCollection 2022 Jul. PMID 36042996